CLINICAL TRIAL: NCT01480804
Title: Identifying and Overcoming Barriers to Diabetes Management in the Elderly: An Intervention Study
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Medha Munshi, Director of Geriactric Diabetes Clinic, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-15
Record Dates: First submitted 2011-11-16; First posted 2011-11-29 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes
Keywords: Barriers; Intervention; Elderly; glycemic control
MeSH Terms: conditions — Diabetes Mellitus | interventions — Methods; Functional Status; Economics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Geriatric diabetes team intervention group (Experimental): The subjects in this group underwent evaluation for barriers to self care by a diabetes educators well versed with age specific barriers. After consideration of patients clinical, functional, and psychosocial background a geriatric diabetes team devised strategy to help patients cope respective barriers. A care manager then implemented the coping strategies by educating patients and caregivers. She also made home visits to assess any safety issues not know to clinic based geriatric team. She helped the patients and caregivers with all aspects of care coordination. Patients in this group received phone contact from care managers as many times as needed over the six month intervention period.
  Interventions: Other: Intervention for age specific barriers to self care
- Attention Control Group (No Intervention): The subjects in the group received similar, in person, contact as the intervention group. An educator, separate from the one involved in the intervention team, called patents in this group for a total of eleven time within the first six months. The phone calls were forces toward general discussion without any diabetes related advice.

INTERVENTIONS:
Other: Intervention for age specific barriers to self care — The intervention included developing strategies to help patients cope with their barriers to self care. The intervention were implemented by care manager over 6 month period in person and by phone calls. During the six to twelve month period subjects did not have any contact with study staff or care manager.
  Other Names: Clinical; Functional; Psychosocial; Economic
  Arms: Geriatric diabetes team intervention group

SUMMARY:
The purpose of this research study is to identify barriers affecting self care in older patients with diabetes and to provide coping strategies for these barriers with help from a care manager (Geriatric Life Specialist) to improve clinical, economical, functional and psychosocial parameters.

DETAILED DESCRIPTION:
This is a study to evaluate whether short term focused intervention by a geriatric diabetes team, with addition of a care manager, to help overcome barriers to diabetes care in older adults will result in improved clinical, functional, and quality of life measures compared to usual care. In addition, we will assess whether the support network formed during intervention by the geriatric diabetes team will empower patients, resulting in long lasting improvement in parameters after intervention is completed. We will also explore whether improved blood glucose control will improve blood circulation in the brain that is compromised in elderly with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and older
* Diagnosis of type 1 or type 2 diabetes
* Seen at Joslin Clinic or Beth Israel Deaconess Medical Center for at least one year
* HbA1c 8% X 2 in past 6 months without fluctuation of more than 0.5% (i.e. stable poor control)
* No major change in medications in past 3 months, e.g. addition of insulin or another hypoglycemic agent

Exclusion Criteria:

* Patients with terminal diseases, e.g. malignancy with life expectancy of 12 months or less
* Patients who live more than 25 miles from Joslin Clinic/ Beth Israel Deaconess Medical Center
* Patients who live in an institutional setting, e.g. nursing home, group home, etc
* Patients who are not able to complete outcome assessments,(e.g. poor vision, diminished mental capacity/severe cognitive decline, unable to speak/read/write English, etc)
* Patients will be excluded from participation in Study Aim 3 if they have a history of orthostatic hypotension, TIA, or vertebral basilar insufficiency

Min Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
change in hemoglobin A1c | 6 and 12 months
  The primary outcome of the study is to measure change in A1c before and after intervention at 6-months and at 12-months

SECONDARY OUTCOMES:
Change in clinical, functional and psycho social tests and questionnaires | 6 and 12 months
  Tests, surveys and questionnaires used during study visits are as follows: Demographic and medical history, hypoglycemia history and calendar, medication adherence survey, modified clock making test, trail making test A and B, verbal fluency test, activities of daily living, instrumental activities of daily living, 6 minute walk test, Tinetti test, geriatric depression scale, problem areas in diabetes assessment, self care inventory, determine nutrition test, social support assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Medha N Munshi, MD, Principal Investigator — Joslin Diabetes Center
Locations (2):
- United States (2):
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts

REFERENCES:
- [Background] Makimattila S, Malmberg-Ceder K, Hakkinen AM, Vuori K, Salonen O, Summanen P, Yki-Jarvinen H, Kaste M, Heikkinen S, Lundbom N, Roine RO. Brain metabolic alterations in patients with type 1 diabetes-hyperglycemia-induced injury. J Cereb Blood Flow Metab. 2004 Dec;24(12):1393-9. doi: 10.1097/01.WCB.0000143700.15489.B2. PMID 15625413
- [Background] Norris SL, Nichols PJ, Caspersen CJ, Glasgow RE, Engelgau MM, Jack L, Isham G, Snyder SR, Carande-Kulis VG, Garfield S, Briss P, McCulloch D. The effectiveness of disease and case management for people with diabetes. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):15-38. doi: 10.1016/s0749-3797(02)00423-3. PMID 11985933
- [Background] Fordyce M, Bardole D, Romer L, Soghikian K, Fireman B. Senior Team Assessment and Referral Program--STAR. J Am Board Fam Pract. 1997 Nov-Dec;10(6):398-406. PMID 9407480
- [Background] Munshi M, Grande L, Hayes M, Ayres D, Suhl E, Capelson R, Lin S, Milberg W, Weinger K. Cognitive dysfunction is associated with poor diabetes control in older adults. Diabetes Care. 2006 Aug;29(8):1794-9. doi: 10.2337/dc06-0506. PMID 16873782
- [Background] Harris MI, Flegal KM, Cowie CC, Eberhardt MS, Goldstein DE, Little RR, Wiedmeyer HM, Byrd-Holt DD. Prevalence of diabetes, impaired fasting glucose, and impaired glucose tolerance in U.S. adults. The Third National Health and Nutrition Examination Survey, 1988-1994. Diabetes Care. 1998 Apr;21(4):518-24. doi: 10.2337/diacare.21.4.518. PMID 9571335
- [Background] Blaum CS, Ofstedal MB, Langa KM, Wray LA. Functional status and health outcomes in older americans with diabetes mellitus. J Am Geriatr Soc. 2003 Jun;51(6):745-53. doi: 10.1046/j.1365-2389.2003.51256.x. PMID 12757559
- [Background] Bertoni AG, Kirk JK, Goff DC Jr, Wagenknecht LE. Excess mortality related to diabetes mellitus in elderly Medicare beneficiaries. Ann Epidemiol. 2004 May;14(5):362-7. doi: 10.1016/j.annepidem.2003.09.004. PMID 15177276
- [Background] Economic consequences of diabetes mellitus in the U.S. in 1997. American Diabetes Association. Diabetes Care. 1998 Feb;21(2):296-309. doi: 10.2337/diacare.21.2.296. PMID 9539999
- [Background] Brown AF, Mangione CM, Saliba D, Sarkisian CA; California Healthcare Foundation/American Geriatrics Society Panel on Improving Care for Elders with Diabetes. Guidelines for improving the care of the older person with diabetes mellitus. J Am Geriatr Soc. 2003 May;51(5 Suppl Guidelines):S265-80. doi: 10.1046/j.1532-5415.51.5s.1.x. No abstract available. PMID 12694461
- [Background] Task Force on Community Preventive Services. Recommendations for healthcare system and self-management education interventions to reduce morbidity and mortality from diabetes. Am J Prev Med. 2002 May;22(4 Suppl):10-4. doi: 10.1016/s0749-3797(02)00422-1. No abstract available. PMID 11985932
- [Background] Baird TA, Parsons MW, Barber PA, Butcher KS, Desmond PM, Tress BM, Colman PG, Jerums G, Chambers BR, Davis SM. The influence of diabetes mellitus and hyperglycaemia on stroke incidence and outcome. J Clin Neurosci. 2002 Nov;9(6):618-26. doi: 10.1054/jocn.2002.1081. PMID 12604269
- [Background] Fulesdi B, Limburg M, Bereczki D, Kaplar M, Molnar C, Kappelmayer J, Neuwirth G, Csiba L. Cerebrovascular reactivity and reserve capacity in type II diabetes mellitus. J Diabetes Complications. 1999 Jul-Aug;13(4):191-9. doi: 10.1016/s1056-8727(99)00044-6. PMID 10616858
- [Background] Griffith DN, Saimbi S, Lewis C, Tolfree S, Betteridge DJ. Abnormal cerebrovascular carbon dioxide reactivity in people with diabetes. Diabet Med. 1987 May-Jun;4(3):217-20. doi: 10.1111/j.1464-5491.1987.tb00865.x. PMID 2956022
- [Background] Kadoi Y, Hinohara H, Kunimoto F, Saito S, Ide M, Hiraoka H, Kawahara F, Goto F. Diabetic patients have an impaired cerebral vasodilatory response to hypercapnia under propofol anesthesia. Stroke. 2003 Oct;34(10):2399-403. doi: 10.1161/01.STR.0000090471.28672.65. Epub 2003 Sep 4. PMID 12958324
- [Background] Jimenez-Bonilla JF, Carril JM, Quirce R, Gomez-Barquin R, Amado JA, Gutierrez-Mendiguchia C. Assessment of cerebral blood flow in diabetic patients with no clinical history of neurological disease. Nucl Med Commun. 1996 Sep;17(9):790-4. doi: 10.1097/00006231-199609000-00009. PMID 8895906
- [Background] MacLeod KM, Gold AE, Ebmeier KP, Hepburn DA, Deary IJ, Goodwin GM, Frier BM. The effects of acute hypoglycemia on relative cerebral blood flow distribution in patients with type I (insulin-dependent) diabetes and impaired hypoglycemia awareness. Metabolism. 1996 Aug;45(8):974-80. doi: 10.1016/s0026-0495(96)90266-8. PMID 8769355
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Bean JF, Kiely DK, Leveille SG, Herman S, Huynh C, Fielding R, Frontera W. The 6-minute walk test in mobility-limited elders: what is being measured? J Gerontol A Biol Sci Med Sci. 2002 Nov;57(11):M751-6. doi: 10.1093/gerona/57.11.m751. PMID 12403805
- [Background] Lord SR, Menz HB. Physiologic, psychologic, and health predictors of 6-minute walk performance in older people. Arch Phys Med Rehabil. 2002 Jul;83(7):907-11. doi: 10.1053/apmr.2002.33227. PMID 12098148
- [Background] Bautmans I, Lambert M, Mets T. The six-minute walk test in community dwelling elderly: influence of health status. BMC Geriatr. 2004 Jul 23;4:6. doi: 10.1186/1471-2318-4-6. PMID 15272934
- [Background] Montorio I, Izal M. The Geriatric Depression Scale: a review of its development and utility. Int Psychogeriatr. 1996 Spring;8(1):103-12. doi: 10.1017/s1041610296002505. PMID 8805091
- [Background] Welch G, Weinger K, Anderson B, Polonsky WH. Responsiveness of the Problem Areas In Diabetes (PAID) questionnaire. Diabet Med. 2003 Jan;20(1):69-72. doi: 10.1046/j.1464-5491.2003.00832.x. PMID 12519323
- [Background] Tiecks FP, Lam AM, Aaslid R, Newell DW. Comparison of static and dynamic cerebral autoregulation measurements. Stroke. 1995 Jun;26(6):1014-9. doi: 10.1161/01.str.26.6.1014. PMID 7762016
- [Background] Panerai RB. Assessment of cerebral pressure autoregulation in humans--a review of measurement methods. Physiol Meas. 1998 Aug;19(3):305-38. doi: 10.1088/0967-3334/19/3/001. PMID 9735883
- [Background] Aaslid R, Newell DW, Stooss R, Sorteberg W, Lindegaard KF. Assessment of cerebral autoregulation dynamics from simultaneous arterial and venous transcranial Doppler recordings in humans. Stroke. 1991 Sep;22(9):1148-54. doi: 10.1161/01.str.22.9.1148. PMID 1926257
- [Background] Zhang R, Zuckerman JH, Giller CA, Levine BD. Transfer function analysis of dynamic cerebral autoregulation in humans. Am J Physiol. 1998 Jan;274(1 Pt 2):H233-41. doi: 10.1152/ajpheart.1998.274.1.h233. PMID 9458872
- [Background] Panerai RB, Dawson SL, Potter JF. Linear and nonlinear analysis of human dynamic cerebral autoregulation. Am J Physiol. 1999 Sep;277(3):H1089-99. doi: 10.1152/ajpheart.1999.277.3.H1089. PMID 10484432
- [Background] Lipsitz LA, Mukai S, Hamner J, Gagnon M, Babikian V. Dynamic regulation of middle cerebral artery blood flow velocity in aging and hypertension. Stroke. 2000 Aug;31(8):1897-903. doi: 10.1161/01.str.31.8.1897. PMID 10926954
- [Background] Benarroch EE, S.P., Low PA, The Valsalva Manuever. In Clinical Autonomic Disroders: Evaluation and Management, L.P. editor, Editor. 1993, Little Brown and company: Boston. p. 209-215.
- [Background] Rutan GH, Hermanson B, Bild DE, Kittner SJ, LaBaw F, Tell GS. Orthostatic hypotension in older adults. The Cardiovascular Health Study. CHS Collaborative Research Group. Hypertension. 1992 Jun;19(6 Pt 1):508-19. doi: 10.1161/01.hyp.19.6.508. PMID 1592445
- [Background] Low, P.A., Laboratory Evaluation of Autonomic Function. In Clinical Autonomic Disorders, P.A. Low, Editor. 1997, LIppincott-Raven: Philadelphia. p. 179-208.
- [Background] Novak V, Chowdhary A, Farrar B, Nagaraja H, Braun J, Kanard R, Novak P, Slivka A. Altered cerebral vasoregulation in hypertension and stroke. Neurology. 2003 May 27;60(10):1657-63. doi: 10.1212/01.wnl.0000068023.14587.06. PMID 12771258
- [Background] Greenfield JC Jr, Rembert JC, Tindall GT. Transient changes in cerebral vascular resistance during the Valsalva maneuver in man. Stroke. 1984 Jan-Feb;15(1):76-9. doi: 10.1161/01.str.15.1.76. PMID 6229907
- [Background] Werner C, Kochs E, Hoffman WE, Blanc IF, Schulte am Esch J. Cerebral blood flow and cerebral blood flow velocity during angiotensin-induced arterial hypertension in dogs. Can J Anaesth. 1993 Aug;40(8):755-60. doi: 10.1007/BF03009772. PMID 8403159
- [Derived] Munshi MN, Segal AR, Suhl E, Ryan C, Sternthal A, Giusti J, Lee Y, Fitzgerald S, Staum E, Bonsignor P, DesRochers L, McCartney R, Weinger K. Assessment of barriers to improve diabetes management in older adults: a randomized controlled study. Diabetes Care. 2013 Mar;36(3):543-9. doi: 10.2337/dc12-1303. Epub 2012 Nov 27. PMID 23193208